CLINICAL TRIAL: NCT05888350
Title: The Value of FeNO, Blood Eosinophils and TIgE in Predicting the Response to Corticosteroid in Patients With Chronic Cough
Brief Title: Biomarkers for Predicting the Response to Inhaled Corticosteroid in Patients With Chronic Cough.
Acronym: CC-ICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Huizhou Third People's Hospital (Unknown); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Nanfang Hospital, Southern Medical University (Other); Shenzhen People's Hospital (Other); SSL Central Hospital of Dongguan City (Unknown); China-Japan Friendship Hospital (Other); Beijing Chao Yang Hospital (Other); Zunyi Medical College (Other); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Second Hospital of Jilin University (Other); Inner Mongolia People's Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Ruijin Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Tongji Hospital (Other); First Hospital of China Medical University (Other); Chongqing Songshan Hospital (Unknown); The First People's Hospital of Yunnan (Other)
Responsible Party: Principal Investigator, Kefang Lai, professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CC-ICS
Record Dates: First submitted 2023-03-27; First posted 2023-06-05 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Cough
Keywords: chronic cough; biomarkers
MeSH Terms: conditions — Cough; Chronic Cough | interventions — Beclomethasone

STUDY DESIGN:
Intervention Model Description: a multi-center, randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foster treatment group (Experimental): Participant inhales Foster (Inhaled Beclometasone Dipropionate and Formoterol Inhalation Aerosol) 1 puff bid for 4 weeks.
  Interventions: Drug: Beclometasone Dipropionate and Formoterol Inhalation Aerosol
- Placebo controlled group (Placebo Comparator): Participant inhales matched placebo 1 puff bid for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Beclometasone Dipropionate and Formoterol Inhalation Aerosol — Inhaled Foster (Beclometasone Dipropionate and Formoterol Inhalation Aerosol) , 1puff, BID, 4weeks
  Arms: Foster treatment group
Drug: Placebo — Inhaled Placebo, 1puff, BID, 4weeks
  Arms: Placebo controlled group

SUMMARY:
To investigate the value of blood eosinophils, FeNO and total IgE in predicting the response to inhaled corticosteroid in patients with chronic cough.

DETAILED DESCRIPTION:
Chronic cough is a frequent complaint in respiratory specialists clinic. CVA, UACS, EB, GERC and AC are common causes of chronic cough, among whom, CVA, EB and AC can be classified as corticosteroid responsive cough.

To recognize the eosinophilic airway inflammation and assess the response of inhaled corticosteroid, induced sputum analysis is the most widely used examination but not all the subjects can provide an suitable sample of sputum for measurements and it's time-consuming.

Recently, blood eosinophils, FeNO and total IgE were detected to be biomarkers of eosinophilic airway inflammation for asthmatics. However, whether can they predict the response to corticosteroid in chronic cough remains uncertain.

The present prospective, multi-center, randomized placebo-controlled study aims to explore the value of blood eosinophils, FeNO and total IgE in predicting the response to inhaled corticosteroid in patients with chronic cough.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years;
2. Coughing lasting ≥ 8 weeks；
3. No abnormality in chest imaging in the past 3 months (or there is abnormality but the investigator judges it not the cause of chronic cough)；
4. FEV1% pred>70%；FEV1/FVC>70%；
5. VAS≥30 in the past 48 hours;
6. Non-smokers or patients smoked less than 10 pack-years;
7. Candidates voluntarily participate in and abide by the relevant regulations of the study, can cooperate with corresponding inspections, follow the follow-up plan, and voluntarily sign written informed consent.

Exclusion Criteria:

1. Patients received inhaled or oral corticosteroids or leukotriene receptor antagonist in previous 4 weeks;
2. Patients with history of upper respiratory tract infection in the past 8 weeks;
3. Patients taking angiotensin-converting enzyme inhibitors in previous 8 weeks;
4. Female subjects who are pregnant, breast-feeding or risk of becoming pregnant during the study;
5. Combined with a definite history of pulmonary diseases such as bronchiectasis, pulmonary interstitial disease, and pulmonary hypertension. Combined with other serious diseases (such as cardiovascular system diseases, metabolic system diseases, immune system diseases, nervous system diseases, etc.) that may affect the normal process of this study;
6. Participating in other drug clinical trial projects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2024-03-02 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
The AUC of blood eosinophils, FeNO and total IgE in predicting the response to inhaled corticosteroid in patients with chronic cough. | the 4th week
  The area under the receiver operating curve (AUC) of blood eosinophils in predicting the response to inhaled corticosteroid in patients with chronic cough.
  The area under the receiver operating curve (AUC) of FeNO in predicting the response to inhaled corticosteroid in patients with chronic cough.
  The area under the receiver operating curve (AUC) of total IgE in predicting the response to inhaled corticosteroid in patients with chronic cough.
The optimal cut-off value of blood eosinophils in cells/μL-1 in predicting the response to inhaled corticosteroid in patients with chronic cough. | the 4th week
  The optimal cut-off value of blood eosinophils in cells/μL-1 in predicting the response to inhaled corticosteroid in patients with chronic cough.
The optimal cut-off value of FeNO in pbb in kU/L in predicting the response to inhaled corticosteroid in patients with chronic cough. | the 4th week
  The optimal cut-off value of FeNO in pbb in predicting the response to inhaled corticosteroid in patients with chronic cough.
The optimal cut-off value of total IgE in kU/L in predicting the response to inhaled corticosteroid in patients with chronic cough. | the 4th week
  The optimal cut-off value of total IgE in kU/L in predicting the response to inhaled corticosteroid in patients with chronic cough.
The sensitivity and specificity in percentage of blood eosinophils, FeNO and total IgE in predicting the response to inhaled corticosteroid in patients with chronic cough. | the 4th week
  The sensitivity and specificity in percentage of blood eosinophils in predicting the response to inhaled corticosteroid in patients with chronic cough.
  The sensitivity and specificity in percentage of FeNO in predicting the response to inhaled corticosteroid in patients with chronic cough.
  The sensitivity and specificity in percentage of total IgE in predicting the response to inhaled corticosteroid in patients with chronic cough.

SECONDARY OUTCOMES:
Clinical characteristics of responders and non-responders | baseline
  Clinical characteristics including gender, age and cough duration would be registered in a specific case report form in baseline.
LCQ change from baseline to the 4th week | the 4th week
  Leicester Cough Questionnaire （LCQ）aims to access the life quality of patients wtih chronic cough, ranging from 19 to 133. Higher scores mean a better outcome.
Cough VAS change from baseline to the 4th week | the 4th week
  Cough visual analogue scale (VAS) aims to access the severity of cough, ranging from 0 to 100mm. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kefang Lai, phD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No